CLINICAL TRIAL: NCT07321925
Title: Thermoacoustic Method for Estimating Liver Fat Fraction - Pilot Study I
Brief Title: Thermoacoustic Method for Estimating Liver Fat Fraction
Status: Recruiting | Type: Observational
Sponsor: Endra Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: ENDRA-CL25-01
Record Dates: First submitted 2025-12-11; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: MASLD/MASH (Metabolic Dysfunction-Associated Steatotic Liver Disease / Metabolic Dysfunction-Associated Steatohepatitis); Fatty Liver Disease, Nonalcoholic
Keywords: Fatty Liver; MASLD; MASH; Thermoacoustic
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Thermoacoustic Enhanced Ultrasound — a novel Thermoacoustic Enhanced imaging device

SUMMARY:
The goal of this study is to use our Thermoacoustic Enhanced Ultrasound device to measure the fat levels in your liver and compare it to the the gold standard MRI PDFF measurements. Participants will have a scan with our device, then they will go have an abdominal MRI completed. The goal is to create a more accessible device to measure liver fat as it is an indicator for overall health and metabolic diseases.

DETAILED DESCRIPTION:
The study will perform thermoacoustic fat measurements for up to 80 participants, over the span of the study. MRI-PDFF sequences will be acquired for participants in the study to establish a true measure of liver fat content, per the MRI gold standard. Determine the correlation between FLIP CID system Fat fraction results and the MRI-PDFF. Determine the accuracy between the fat measures obtained by the FLIP CID system participants who received a quantitative MRI. The following additional parameters will be evaluated endpoints: Sensitivity, Specificity ,Positive and negative predictive value (PPV, NPV) and The area under the ROC curve for the detection of liver fat abnormalities

ELIGIBILITY:
Inclusion Criteria:

* Study participants are 18 or older.
* Able to understand, read, and provide written informed consent in English.
* Able to tolerate both ultrasound and MRI examinations.
* Able to lie flat, or on their side, for 20 minutes and pause breathing for up to 10 seconds.

Exclusion Criteria:

* Metal or electronic implants, including, but not limited to: pacemakers, metal clips, drug delivery pumps, hip implants, and neural stimulation devices, contraindicates for MRI.
* Known pregnancy the day of consent or becoming pregnant during study participation based on start date of last menstrual period).
* Liver diseases other than MASLD/MASH/fibrosis including, but not limited to:
* Cirrhosis
* Hepatocellular carcinoma
* Ascites
* Patients with broken, or injured skin, in the right upper abdominal quadrant.
* Body habitus, or anatomical variation, where the liver capsule is not accessible with ultrasound through the patient's right intercostal imaging window used in conventional ultrasound liver imaging.
* BMI greater than 50 kg/m2
* Patients with subcutaneous fat at measurement location less than or equal to 6mm.
* Patients with a missing liver lobe.
* Patients with peri-hepatic fat in the measurement location.
* Patients with focal liver lesions or anatomical structures in the measurement location, as detected by ultrasound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study Participants will be from the local general population with focus on potential study participants with known, or clinically suspected, elevated fatty liver
Sampling Method: Non-Probability Sample
Enrollment: 49 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between Thermoacoustic Fat Fraction (TAFF) and the MRI-PDFF | From enrollment until the statistical analysis is reviewed, typically 2 weeks after last MRI data is received.
  The correlation between TAFF and the MRI-PDFF, will be conducted using the calculation of the cumulative distribution of the correlation coefficient as derived by Guenther

CONTACTS AND LOCATIONS:
Locations (1):
- ENDRA Life Sciences, Ann Arbor, Michigan, United States